CLINICAL TRIAL: NCT00578630
Title: Interindividual Genetic Variability as a Determinant of Chemotherapy Toxicity and Response in Pediatric Oncology/Bone Marrow Transplantation Patients
Brief Title: Interindividual Genetic Variability as a Determinant of Chemotherapy Toxicity and Response in Pediatric Bone Marrow Transplantation Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Cancer Society, Inc. (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 03-123; NCI CA 83132
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Neoplasms
Keywords: pediatric tumors; genetic test development; All Pediatric patients with a histologically proven tumor.
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood and buccal swab

GROUPS / COHORTS (1):
- 1: All Pediatric Oncology and Bone Marrow Transplantation Service patients with a histologically proven tumor for whom there is an intent to treat with chemotherapy
  Interventions: Other: buccal swabs and obtaining peripheral blood

INTERVENTIONS:
Other: buccal swabs and obtaining peripheral blood — will be the collection of normal cells and assessments of toxicity following chemotherapy at routine clinic visits.

SUMMARY:
The purpose of this study is to develop tests that will allow us to determine who will react differently to the drugs used to treat cancer. We also want to see who will react differently with preparing for a bone marrow transplant.

DETAILED DESCRIPTION:
The title of this study is interindividual genetic variability as a determinant of chemotherapy toxicity and response in pediatric oncology/bone marrow transplantation patients. We will collect blood from pediatric oncology/bone marrow transplantation patients who are going to receive chemotherapy in order to assess several defined genetic polymorphisms that may be involved in chemotherapy toxicity and response. The polymorphisms will be assessed on normal mononuclear cells by a combination of techniques. We will determine whether these polymorphisms occur in pediatric oncology/bone marrow transplantation patients and their correlation with different clinical features during and following therapy including toxicity and response. The presence or absence of polymorphisms will be correlated with patient outcome and tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

* All Pediatric Oncology and Bone Marrow Transplantation Service patients with a histologically proven tumor for whom there is an intent to treat with chemotherapy are eligible for participation in this study. The patient does not need to be newly diagnosed for enrollment on this protocol.
* All patients or their guardians must provide written informed consent. Minors will be required to provide assent.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Pediatric Oncology and Bone Marrow Transplantation Service patients with a histologically proven tumor for whom there is an intent to treat with chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2003-10-14 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
To determine if genetic polymorphisms are associated with the presence and extent of chemotherapy related toxicity in pediatric bone marrow transplantation patients and the response and outcome of these patients. | 12 months

SECONDARY OUTCOMES:
To determine if the presence of genetic polymorphisms are associated with the response and outcome of pediatric oncology/bone marrow transplantation patients. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Meyers, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org